CLINICAL TRIAL: NCT03065972
Title: A Randomized Controlled Comparative Study on Efficacy and Cost-effectiveness of Autologous Arteriovenous Fistulas Versus Hemodialysis Access Grafts in Elderly Patients
Brief Title: Hemodialysis in the Elderly (70yrs & Older)
Acronym: ELDERLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: E. Peden, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, E. Peden, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013220
Record Dates: First submitted 2016-07-15; First posted 2017-02-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Kidney Disease; Kidney Failure; Chronic Kidney Disease
Keywords: kidney disease; vascular access; graft; fistula; hemodialysis; dialysis
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Renal Insufficiency, Chronic; Fistula | interventions — Portacaval Shunt, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical fistula creation from patient's anatomy (Active Comparator): Patients randomized to surgical arteriovenous fistula will have a fistula surgically created from their anatomy to be used for hemodialysis access.
  Interventions: Procedure: Surgical fistula creation from patient's anatomy
- Surgical graft implant (Active Comparator): Patients randomized to surgical graft, will have a commercially available graft surgically implanted to be used for hemodialysis access.
  Interventions: Procedure: Surgical fistula creation from patient's anatomy; Device: Surgical Graft implant

INTERVENTIONS:
Procedure: Surgical fistula creation from patient's anatomy — Patient will be randomized via computer system, to receive the fistula or graft. If fistula, surgeon creates fistula for hemodialysis access from patient's anatomy.
  Other Names: Fistula
Device: Surgical Graft implant — Patient will be randomized via computer system, to receive the fistula or graft. If graft, surgeon implants hemodialysis access using an FDA approved graft.
  Other Names: FDA approved graft (various manufacturers)
  Arms: Surgical graft implant

SUMMARY:
This will be a prospective, single institution, parallel-group, single-blinded, randomized-controlled, two-arm, effectiveness study comparing autologous arteriovenous fistula versus hemodialysis access grafts in the elderly. The target sample size will include enrollment of 270 patients over a period of 5 years. The creation of an autologous arteriovenous fistula or placement of a hemodialysis access graft constitutes the two arms of the study.

DETAILED DESCRIPTION:
This will be a prospective, single institution, parallel-group, single-blinded, randomized-controlled, two-arm, effectiveness study comparing autologous arteriovenous fistula versus hemodialysis access grafts in the elderly. The target sample size will include enrollment of 270 patients over a period of 5 years. The creation of an autologous arteriovenous fistula or placement of a hemodialysis access graft constitutes the two arms of the study.

Following the access creation the patients will be followed-up as per the standard and study protocol for a period of 2 years from the time of access creation.

The investigators will use block randomization to achieve a patient allocation ratio of 1:1, using varying blocks of sizes 4 and 6 in a random order as per a web-based/computer generated system maintained as a block randomization sequence/list concealed from the blinded clinical and trial research team until the end of trial. Patients will be randomly allocated based on this permuted sequence to either of the two intervention groups.

Masking will be performed and shall involve blinding of the patients participating in the trial. The research assistants involved with consenting, enrolling, data collection and follow-up, and the statistician analyzing the outcome measures will be blinded to the group assignment. The operating surgeon shall be blinded to the allocation process until the time of access creation following which the knowledge regarding the type of access creation by the surgeon is inevitable. All patients will be consented and their study related details including history, physical evaluations, diagnostic tests, etc., will be entered on a case report form and maintained on a web-based database. The patients will be followed-up for a period of 2 years from the time of initial access creation until the access is abandoned or rendered nonfunctional until the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥70 years of all ethnicities, and;
* Have vascular anatomy amenable to arteriovenous fistula creation, and;
* Diagnosed with End-stage Renal Disease stage 4 (GFR 15-29 ml/min 1.73m2) or stage 5 (GFR <15ml/min 1.73m2) as per the National Kidney Foundation guidelines needing vascular access for hemodialysis; or,
* Currently undergoing hemodialysis with a failure of previous access; or,
* Expected to undergo hemodialysis within 6 months of presentation.

Exclusion Criteria:

* Unable or refuse to abide with follow-up; or,
* Known hypercoagulability syndrome or a bleeding disorder; or,
* Intraoperative decision was made in favor of fistula instead of graft; or,
* Active infections; or,
* Evidence or suspicion of central vein stenosis but shall be included if a central vein catheter or pacemaker is implanted as long as the patient had a venogram within past 6 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-01-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Analyze hemodialysis (HD) access creation, arteriovenous (AV) fistula vs Graft, in elderly patients. | 12 months
  Assess frequency of HD access use, abandonment, and patency at 12 months post-procedure. We will communicate with the patient every month from date of surgery until 12 months to complete questionnaires to determine access use and patency for their study related access creation
Functional cumulative patency rate at 12 months | 12 months
  Functional refers to the availability of the access for hemofiltration. Primary patency refers to the successful use of a vascular access for hemodialysis without any surgical or endovascular intervention

SECONDARY OUTCOMES:
Using Disease Outcomes Quality Initiative quality of life tool to evaluate and compare the overall improvement in outcome with respect to morbidity in the 2 years post fistula/graft procedure | 2 years
  Using Disease Outcomes Quality Initiative quality of life tool
To compare and analyze the estimated costs with both types of hemodialysis interventions and their postoperative outcomes. | 2 years
  Analysis of hospital bills to compare the costs with both types of hemodialysis interventions
Using Disease Outcomes Quality Initiative quality of life tool to evaluate and compare the overall improvement in outcome with respect to mortality in the 2 years post fistula/graft procedure | 2 years
  Using Disease Outcomes Quality Initiative quality of life tool
Using Disease Outcomes Quality Initiative quality of life tool to evaluate and compare the overall improvement in outcome with respect to patient's quality of life in the 2 years post fistula/graft procedure | 2 years
  Using Disease Outcomes Quality Initiative quality of life tool

CONTACTS AND LOCATIONS:
Overall Officials: Eric K Peden, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Investigators plan to write a manuscript once all the participant information has been compiled.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Available for 5 years upon study completion
Access Criteria: After publication of results, de-identified participant data can be made available upon reasonable request to the Primary Investigator